CLINICAL TRIAL: NCT05684874
Title: Neoadjuvant Radiotherapy of Soft Tissue Sarcomas of Limbs and Trunk : Interest of Multiparametric Quantitative MRI for Response Assessment and Per-treatment Progression Prediction
Brief Title: Multiparametric Quantitative MRI and Response to Neoadjuvant Radiotherapy for Soft-tissue Sarcoma
Acronym: SarQuantIRM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ET22-301
Record Dates: First submitted 2022-11-24; First posted 2023-01-13 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Soft Tissue Sarcoma; Adult Soft Tissue Sarcoma; Resectable Soft Tissue Sarcoma
Keywords: Oncology; Soft Tissue Sarcoma; Multiparametric quantitative MRI; Neoadjuvant radiotherapy; Limbs and trunk; Remnographic characteristics; Tumor resection; Anatomopathological response; Predictive biomarkers; Complete pathological response; Change in tumor volume; Adults; Resectable
MeSH Terms: conditions — Sarcoma; Neoplasms; Pathologic Complete Response | interventions — Transurethral Resection of Bladder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre- and post- radiotherapy multiparametric quantitative MRI (Experimental): Patients with STS of the limbs and trunk will be accrued during the initial radiotherapy consultation radiotherapy (prior to receiving radiotherapy).
  Two quantitative multiparametric MRI will be performed. The first one will be acquired less than 14 days before the dosimetric scan, the second one 4 to 6 weeks after the end of the radiotherapy.
  A tumor resection will be performed 6 to 8 weeks post-RT and an anatomopathological observation of the surgical specimen will be performed.
  Interventions: Radiation: Neoadjuvant RT; Other: Pre-radiotherapy mpMRI; Other: Post-radiotherapy mpMRI; Procedure: Tumor resection

INTERVENTIONS:
Radiation: Neoadjuvant RT — Dosimetric CT scan with contrast injection for treatment planning. Radiation therapy at a dose of 50Gy in 25 fractions, 5 fractions per week. Daily pre-treatment positioning tomographic imaging (either high energy (MVCT) or cone beam computed tomography (CBCT)).
  Delineation of the tumor volume and evaluation of its evolution. In case of change of volume and if medically relevant, new dosimetric scan and collection of the tumor volume.
Other: Pre-radiotherapy mpMRI — Performed less than 14 days before the dosimetric scan. Conventional morphological T1-weighted, T2-weighted, and T1-weighted imaging sequences after injection of contrast agent.
  Quantitative imaging sequences including multiple b-value diffusion imaging. Chemical shift sensitized sequences.
Other: Post-radiotherapy mpMRI — Performed 4 to 6 weeks after the end of the radiotherapy. Conventional morphological T1-weighted, T2-weighted, and T1-weighted imaging sequences after injection of contrast agent.
  Quantitative imaging sequences including multiple b-value diffusion imaging. Chemical shift sensitized sequences.
Procedure: Tumor resection — Performed 6 to 8 weeks after the end of radiotherapy. An anatomopathological observation of the surgical specimen will be performed.

SUMMARY:
This trial is a prospective, monocentric, with minimal risks and constraints study, conducted in patients with Soft Tissue Sarcoma (STS) of the limbs and trunk with indication for neoadjuvant radiotherapy (RT).

Patients will be treated by neoadjuvant RT and will have a pre-RT and a post-RT multiparametric quantitative Magnetic Resonance Imaging (MRI).

A tumor resection will be performed 6 to 8 weeks post-RT and an anatomopathological observation of the surgical specimen will be performed.

This study will allow to describe the initial remnographic characteristics and their evolution after neoadjuvant RT using quantitative multiparametric MRI (mpMRI).

DETAILED DESCRIPTION:
This study is prospective, monocentric and with minimal risks and constraints.

Patients with STS of the limbs and trunk will be accrued during the initial radiotherapy consultation radiotherapy (prior to receiving radiotherapy).

Two quantitative multiparametric MRI will be performed. The first one will be acquired less than 14 days before the dosimetric scan, the second one 4 to 6 weeks after the end of the radiotherapy.

This study will allow to describe the initial remnographic characteristics and their evolution after neoadjuvant RT using quantitative multiparametric MRI.

STATISTICAL ANALYSIS

Patients will be systematically recruited from December 2022 to August 2023, i.e. a potential of approximately 20-30 patients.

Analysis conventions:

Categorical variables will be expressed as numbers and percentages, and continuous variables as median (minimum-maximum). The normality of the distributions of the quantitative MRI data will be assessed by a Shapiro-Wilk test. A p-value <0.05 will be considered significant with two-tailed tests. No imputation will be performed in case of missing data. Statistical analyses will be performed using R software (R Foundation for Statistical Computing, Vienna, Austria).

Analysis of the primary endpoint:

The remnographic parameters observed pre- and post-radiotherapy will be described, both qualitatively in T1 weighting, T2 with and without fat saturation, T1 with gadolinium injection, and quantitatively in Chemical Shift-Encoded (CSE) MRI sequence, T2 mapping and multi-echo gradient diffusion.

Analysis of secondary endpoints:

The clinico-remnographic data of the groups with and without complete pathological response will be compared using Student's t test, Wilcoxon test, Chi2 test or Fisher's exact test when appropriate.

ROC curves will be generated to assess the performance of the remnographic parameters in predicting pathological complete response as well as in predicting per-treatment progression via the use of the area under the Receiver Operator Characteristic (ROC) curve (AUC). The Youden index will be used to identify the optimal threshold.

Univariate and multivariate logistic regressions will be performed to assess the clinico-remnographic parameters predictive of complete pathological response as well as those predictive of per-treatment progression.

A Student's t test or a Wilcoxon test will be performed to evaluate the correlation between pre-radiotherapy remnographic parameters and the percentage of variation in tumour volume during treatment, as well as between pre-operative remnographic parameters and the percentage of necrosis on anatomopathological examination of the surgical specimen.

DATA ENTRY, DATA MANAGEMENT AND STUDY MONITORING

Data generated within the framework of the study will be entered, for each patient, by the investigator of the centre (or a person designated by delegation) on an Excel file in a secure location on the internal network of the Centre Léon Bérard.

Only New Safety Issues occurring in the course of the study will be reported. A New Safety Issue is defined as any new data that could lead to reevaluate the ratio between the benefits and the risks of the research, or that could be sufficiently important to consider modifications of the research documents, the research management or, to suspend, to interrupt or to modify the protocol of the research or of similar researches. The Sponsor should report without delay any New Safety Issue, as well as any safety measures to be proposed, discussed with the principal investigator, to the Ethics Committee and the principal investigators. Relevant follow-up information will be provided within a further 8 days.

The sponsor will assist the investigator in the conduct of the study in accordance with the study protocol, Good Clinical Practice and the regulations in force.

At regular intervals during the study, a representative of the coordinating centre may contact the investigating team in order to control the progress of the project, investigator and patient compliance with the protocol and to identify any potential problem in the study.

ELIGIBILITY:
INCLUSION CRITERIA :

* Patients 18 years of age or older;
* Documented histologic diagnosis of soft tissue sarcoma of the limbs or trunk;
* Validated indication for neoadjuvant radiotherapy, planned in the radiotherapy department of the Centre Léon Bérard;
* No contraindication to Magnetic Resonance Imaging,
* Signed informed consent;
* Affiliation with a social security system or beneficiary of such a system.

EXCLUSION CRITERIA :

* Tumor considered as unresectable or patient considered as non-operable;
* Desmoid tumor or dermatofibrosarcoma protuberans due to intermediate malignancy;
* Rhabdomyosarcoma due to a different therapeutic management;
* Multi-metastatic disease;
* Pregnant or lactating woman,
* Patient under guardianship, curatorship or deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Maximum axial dimension | Pre-radiotherapy mpMRI performed within 14 days before the dosimetric scan. Post-radiotherapy mpMRI performed 4 to 6 weeks after radiation therapy completion.
  Evolution of the maximum axial dimension (mm) after neoadjuvant radiotherapy, obtained with quantitative multiparametric MRI
Volume of the region of interest (ROI) | Pre-radiotherapy mpMRI performed within 14 days before the dosimetric scan. Post-radiotherapy mpMRI performed 4 to 6 weeks after radiation therapy completion.
  Evolution of the volume of the region of interest (ROI) (mm3) after neoadjuvant radiotherapy, obtained with quantitative multiparametric MRI
Minimum, maximum, mean, median, 10th, 25th, 75th and 90th percentile values of free diffusion (D) and microperfusion-related diffusion (D*). | Pre-radiotherapy mpMRI performed within 14 days before the dosimetric scan. Post-radiotherapy mpMRI performed 4 to 6 weeks after radiation therapy completion.
  Evolution of the minimum, maximum, mean, median, 10th, 25th, 75th and 90th percentile values of free diffusion (D) and microperfusion-related diffusion (D*) (mm2/s) after neoadjuvant radiotherapy, obtained with quantitative multiparametric MRI
Fraction of perfusion (f) | Pre-radiotherapy mpMRI performed within 14 days before the dosimetric scan. Post-radiotherapy mpMRI performed 4 to 6 weeks after radiation therapy completion.
  Evolution of the fraction of perfusion (f) after neoadjuvant radiotherapy, obtained with quantitative multiparametric MRI

SECONDARY OUTCOMES:
Predictive biomarker of complete pathological response in pre-radiotherapy mpMRI | Pre-radiotherapy mpMRI performed within 14 days before the dosimetric scan. Surgery performed 6 to 8 weeks after radiation therapy completion.
  ROC curves will be generated to evaluate the performance of remnographic parameters for the prediction of complete pathological response using the area under the ROC curve (AUC).

OTHER OUTCOMES:
Predictive biomarkers of risk factors for tumor progression in pre-radiotherapy mpMRI | Pre-radiotherapy mpMRI performed within 14 days before the dosimetric scan. 5 weeks of daily image guided radiotherapy.
  ROC curves will be generated to evaluate the performance of remnographic parameters for the prediction of per-treatment progression using the area under the ROC curve (AUC).
Remnographic data and anatomopathological specimen results | 4 to 6 weeks after radiation therapy completion (remnographic data), and 6 to 8 weeks after radiation therapy completion (anatomopathological specimen results).
  Qualitative geographic correlation between post-radiotherapy remnographic data and pathological observation of necrosis, fibrosis and perennial cell areas.

CONTACTS AND LOCATIONS:
Overall Officials: Benoît ALLIGNET, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Léon Bérard, Lyon, Rhône, France